CLINICAL TRIAL: NCT02563587
Title: Efficacy of the Spontaneous Laughter on Postoperative Pain and Anxiety in Children. A Randomized Controlled Trial
Brief Title: Efficacy of Spontaneous Laughter in the Postoperative Treatment of Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Naval de Alta Especialidad - Escuela Medico Naval (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HGNAE-02; pecm830703 (Registry Identifier: Magda Ruth Pérez Cervantes)
Record Dates: First submitted 2015-09-11; First posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Pain
Keywords: Laughter; children; postoperative; pain; anxiety; cortisol
MeSH Terms: conditions — Pain; Laughter; Anxiety Disorders | interventions — Laughter Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group LT-CT (Experimental): Laughter therapy with conventional treatment
  Interventions: Other: Laughter therapy
- Group AW-CT (Placebo Comparator): Accompaniment without causing the laughter of children more conventional treatment
  Interventions: Other: Accompaniment without causing the laughter of children.
- Group CT (Sham Comparator): Conventional treatment only
  Interventions: Drug: Conventional treatment

INTERVENTIONS:
Other: Laughter therapy — Laughter therapy sessions will begin as soon as / after that the complete anesthesia recovery, then we could start with two interventions, each of them in morning and during the afternoon will be held until their discharge lasting 30 minutes per each one, these sessions will be held in the service pediatric hospital by trained personnel in laughter therapy, which will be implemented through hospital clowns.
  Other Names: Group LT-CT
  Arms: Group LT-CT
Other: Accompaniment without causing the laughter of children. — The interventions will be carried out by means of reading stories and own stories for the age. These sessions will begin subsequent to the full recovery of the anesthesia, and then two interventions per day, in the morning and evening, with duration of 30 minutes, until the time of his discharge, these sessions will take place in the service of Hospital pediatrics by the resident in charge.
  Other Names: Group AW-CT
  Arms: Group AW-CT
Drug: Conventional treatment — Conventional treatment involves handling analgesic with non-steroidal anti-inflammatory drugs (paracetaol, metamizol and ketorolac) as prescribed by the doctor surgeon treating, which starts immediately in the postoperative period.
  Other Names: Group CT
  Arms: Group CT

SUMMARY:
The purpose of this study is to determine the efficacy of laughter therapy in children to improve postoperative, evaluating the intensity of postoperative pain, anxiety and hospital stay.

DETAILED DESCRIPTION:
The therapeutic efficacy of laughter is supported in several research which have shown to have preventive and therapeutic effects that contribute to a better quality of life. In addition, laughter can optimize strategies to increase pain tolerance and combat stress, reducing the negative impact such as increased blood pressure, decreases simultaneously perfusion of organs not needed for the motor function, increased metabolism rates cell with increased serum cortisol and increased risk of infections. Nevertheless the upswing in research on these effects, there is still a necessity to have evidence-based medicine as most of the available studies are limited by various problems such as lack of objectivity in the assessment and measurement, distinction between laughter and mood, establishment dosing therapies (frequency and time).

The aim of our study is to determine the efficacy of spontaneous laughter in children to improve postoperative pain, anxiety and length of hospital stay.

Methods: A controlled, randomized, open label trial with an experimental group exposed to the conventional pain treatment with laughter therapy; 2 control group, a group with accompaniment without causing the laughter of children to control the effect of a companion instead of the clown and a conventional treatment group to contrast with experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients between 6 and 14
* I hospitalized with uncomplicated surgical procedure
* Minimum period of hospitalization of 48 hours
* Patients with informed consent letter signed by parents or guardians
* In patients older than 10 years, a letter of agreement

Exclusion Criteria:

* Endocrinopathies carriers, cancer, abnormalities of central nervous system immune disorders patients.
* Patients treated with both topical and systemic steroids

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain level | 48 hours after surgery
  Pain level measurement at 48 hours determined by the visual analogue scale (Range: 0-10 cm)

SECONDARY OUTCOMES:
Postoperative anxiety level | 48 hours after surgery
  Postoperative anxiety level determined by STAIC (State Trait Anxiety Inventory Children) (Range: 10-40 points)
Postoperative urinary cortisol level | 48 hours after surgery
  Postoperative stress level determined by urinary cortisol (μg/dl)
Postoperative heart rate | 48 hours after surgery
  Postoperative heart rate (beat per minute)
Postoperative respiratory rates | 48 hours after surgery
  Postoperative breathing frequency (breath per minute)
Postoperative systolic blood pressure | 48 hours after surgery
  Postoperative systolic blood pressure (mmHg)
Postoperative diastolic blood pressure | 48 hours after surgery
  Postoperative diastolic blood pressure (mmHg)
Postoperative oxygen saturation | 48 hours after surgery
  Postoperative oxygen saturation (%)
Length of hospital stay | 168 hours after surgery
  Postoperative hospital stay length (hours)

CONTACTS AND LOCATIONS:
Overall Officials: Magda Ruth Pérez Cervantes, Pediatrician, Principal Investigator — Secretaria de Marina
Locations (1):
- Hospital General Naval de Alta Especialidad, Mexico City, Mexico City, Mexico

REFERENCES:
- [Result] Guzmán SV, Torres HJ, Plascencia HA, Castellanos MJ, Quintanilla MR. Cultura hospitalaria y el proceso narrativo en el niño enfermo. Estudio sobre las Culturas Contemporáneas. 2011 jul; XVII (33): 23-44
- [Result] González ML, Gallardo DE. Calidad de la atención médica: La diferencia entre la vida o la muerte. Revista digital universitaria UNAM. 2012 Ago; 13 (8)
- [Result] Hernandez PE, Rabadan RJ. Hospitalization, a break in the child´s life. Educational attention in infantile hospitalized population. Perspectiva Educacional. 2013 Ene; 52 (1):167-181
- [Result] Meisel V, Chellew K, Ponsell E, Ferreira A, Bordas L, Garcia-Banda G. [The effect of "hospital clowns" on distress and maladaptive behaviours of children who are undergoing minor surgery]. Psicothema. 2009 Nov;21(4):604-9. Spanish. PMID 19861106
- [Result] Griffin GD, Charron D, Al-Daccak R. Post-traumatic stress disorder: revisiting adrenergics, glucocorticoids, immune system effects and homeostasis. Clin Transl Immunology. 2014 Nov 14;3(11):e27. doi: 10.1038/cti.2014.26. eCollection 2014 Nov. PMID 25505957
- [Result] Guyton y Hall. Tratado de Fisiología médica. Editorial ELSEVIER. 2011; 12: 1052-1055
- [Result] Heden LE, von Essen L, Ljungman G. Effect of morphine in needle procedures in children with cancer. Eur J Pain. 2011 Nov;15(10):1056-60. doi: 10.1016/j.ejpain.2011.05.010. Epub 2011 Jun 15. PMID 21680210
- [Result] Brasher C, Gafsous B, Dugue S, Thiollier A, Kinderf J, Nivoche Y, Grace R, Dahmani S. Postoperative pain management in children and infants: an update. Paediatr Drugs. 2014 Apr;16(2):129-40. doi: 10.1007/s40272-013-0062-0. PMID 24407716
- [Result] Montero-Homs J. [Nocioceptive pain, neuropathic pain and pain memory]. Neurologia. 2009 Jul-Aug;24(6):419-22. Spanish. PMID 19798608
- [Result] Finley GA, Kristjansdottir O, Forgeron PA. Cultural influences on the assessment of children's pain. Pain Res Manag. 2009 Jan-Feb;14(1):33-7. doi: 10.1155/2009/763031. PMID 19262914
- [Result] Noel M, Chambers CT, McGrath PJ, Klein RM, Stewart SH. The role of state anxiety in children's memories for pain. J Pediatr Psychol. 2012 Jun;37(5):567-79. doi: 10.1093/jpepsy/jss006. Epub 2012 Feb 23. PMID 22362922
- [Result] Christian R, Ramos J, Susanibar C, Balarezo G. Laugh Therapy: A new field for healthcare professionals. Rev. Soc. Per. Med. Inter. 2004; 17(2)
- [Result] Gendry S. Certified Laughter Yoga Teacher Workbook. American School of Laughter Yoga. 2013
- [Result] Nasr SJ. No laughing matter: laughter is good psychiatric medicine. A case report. Current Psychiatry. 2013; 12(8): 20-25
- [Result] Amez AJ, Díaz PM. Manejo del dolor en odontopediatría. Rev Estomatol Herediana. 2010; 20(3):166-171
- [Result] Takeda M, Hashimoto R, Kudo T, Okochi M, Tagami S, Morihara T, Sadick G, Tanaka T. Laughter and humor as complementary and alternative medicines for dementia patients. BMC Complement Altern Med. 2010 Jun 18;10:28. doi: 10.1186/1472-6882-10-28. PMID 20565815
- [Result] Woodbury-Farina MA, Antongiorgi JL. Humor. Psychiatr Clin North Am. 2014 Dec;37(4):561-78. doi: 10.1016/j.psc.2014.08.006. Epub 2014 Nov 25. PMID 25455066
- [Result] Pearce JM. Some neurological aspects of laughter. Eur Neurol. 2004;52(3):169-71. doi: 10.1159/000081857. Epub 2004 Nov 2. PMID 15528918
- [Result] Rodríguez AC, Magallanes MA, Estañol VB, Tovar VJ, Valencia FM. Aspectos neurológicos y neurofisiología de la risa. Arch Neurocien INNN. 2000; 5(1): 43-49
- [Result] Lancheros GE, Tovar VJ, Rojas BC. Laughter and health: therapeutic approaches. Med UNAB. 2011 jul; 14(1): 69-75
- [Result] Kimata H. Effect of humor on allergen-induced wheal reactions. JAMA. 2001 Feb 14;285(6):738. doi: 10.1001/jama.285.6.738. No abstract available. PMID 11176910
- [Result] Mora Ripoll R, Garcia Rodera MC. [Therapeutical value of laughter in medicine]. Med Clin (Barc). 2008 Nov 22;131(18):694-8. doi: 10.1157/13129114. No abstract available. Spanish. PMID 19087828
- [Result] Vagnoli L, Caprilli S, Robiglio A, Messeri A. Clown doctors as a treatment for preoperative anxiety in children: a randomized, prospective study. Pediatrics. 2005 Oct;116(4):e563-7. doi: 10.1542/peds.2005-0466. PMID 16199685
- [Result] Bennett MP, Zeller JM, Rosenberg L, McCann J. The effect of mirthful laughter on stress and natural killer cell activity. Altern Ther Health Med. 2003 Mar-Apr;9(2):38-45. PMID 12652882
- [Result] Mifflin KA, Hackmann T, Chorney JM. Streamed video clips to reduce anxiety in children during inhaled induction of anesthesia. Anesth Analg. 2012 Nov;115(5):1162-7. doi: 10.1213/ANE.0b013e31824d5224. Epub 2012 Oct 9. PMID 23051880
- [Result] Yip P, Middleton P, Cyna AM, Carlyle AV. Non-pharmacological interventions for assisting the induction of anaesthesia in children. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD006447. doi: 10.1002/14651858.CD006447.pub2. PMID 19588390
- [Result] Fernandes SC, Arriaga P. The effects of clown intervention on worries and emotional responses in children undergoing surgery. J Health Psychol. 2010 Apr;15(3):405-15. doi: 10.1177/1359105309350231. PMID 20348361
- [Result] Chang C, Tsai G, Hsieh CJ. Psychological, immunological and physiological effects of a Laughing Qigong Program (LQP) on adolescents. Complement Ther Med. 2013 Dec;21(6):660-8. doi: 10.1016/j.ctim.2013.09.004. Epub 2013 Sep 13. PMID 24280475
- [Result] Villamil M, Quintero A, Henao E, Cardona JL. Terapia de la risa en un grupo de mujeres adultas. Rev. Fac. Nac. Salud Pública 2013;31(2):202-208
- [Result] Sakai Y, Takayanagi K, Ohno M, Inose R, Fujiwara H. A trial of improvement of immunity in cancer patients by laughter therapy. Jpn Hosp. 2013 Jul;(32):53-9. PMID 23984543